CLINICAL TRIAL: NCT06173219
Title: A Prospective Clinical Trial Evaluating the Safety and Efficacy of Radiotherapy Combined with Immunotherapy in Advanced Refractory Solid Malignancies After Standard Treatment Failure/drug Resistance.
Brief Title: Safety and Efficacy of Radiotherapy Combined with Immunotherapy for Advanced Malignant Tumors.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Guangying Zhu, chief physician, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-ZF-63
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumor; standard treatment failure; radiotherapy; immunotherapy
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): The subjects will receive the combination therapy of SBRT, LDRT, PD-1/L1 inhibitor and GMCSF. The specific treatment regimen is as follows: (1) SBRT 8Gy×3f, (2) LDRT 2Gy ×3f, PD-1/L1 inhibitor, periodically, until the disease progresses or intolerable toxic side effects, (4) GM-CSF, 200ug/QD, subcutaneous injection, the first course of treatment for 7 days.
  Interventions: Combination Product: Radiotherapy combined with immunotherapy

INTERVENTIONS:
Combination Product: Radiotherapy combined with immunotherapy — (1) SBRT 8Gy×3f, (2) LDRT 2Gy ×3f, PD-1/L1 inhibitor, periodically, until the disease progresses or intolerable toxic side effects, (4) GM-CSF, 200ug/QD, subcutaneous injection, the first course of treatment for 7 days.

SUMMARY:
The goal of this clinical trial is to find a new radioimmunotherapy regimen for advanced malignancies with multiple metastatic after standard treatment failure/drug resistance. The main questions it aims to answer is: the safety and efficacy of the new regimen for advanced multiple metastatic solid tumors standard treatment failure/drug resistance, and explore the impact on immune function. Participants will receive the combination of radiotherapy and immunotherapy.

DETAILED DESCRIPTION:
More effective treatment regimens remain to be explored for advanced malignancies with multiple metastatic after standard treatment failure/drug resistance. The combination of radiotherapy and immunotherapy is considered to be a promising therapeutic strategy. Studies showed the efficacy of PRaG (PD-1 inhibitor, Radiotherapy and GM-CSF) treatment and stereotactic radiotherapy (SBRT) combined with low-dose radiotherapy (LDRT) for advanced tumors. Therefore, the investigators designed a new radioimmunotherapy regimen, including SBRT, LDRT , PD-1/PD-L1 inhibitor, and GM-CSF. This study aimed to evaluate the safety and efficacy of the new regimen for advanced multiple metastatic solid tumors standard treatment failure/drug resistance, and explore the impact on immune function.

ELIGIBILITY:
Inclusion Criteria:

1. advanced malignant solid tumors with multiple metastases or relapses, with pathological diagnosis or medical record;
2. disease progression or recurrence after standard treatment, or unsuitable/intolerable for standard treatment, or rejection of standard treatment due to personal willingness;
3. patients with disease progression or drug resistance after previous immunotherapy are allowed to be included; a history of radiotherapy in the LDRT area or other sites is allowed to be included, provided that there are no residual toxic effects;
4. at least ≥1 lesion suitable for SBRT, and ≥1 lesion suitable for LDRT, and the above lesions must be measured;
5. no contraindications to radiotherapy;
6. Eastern Cooperative Oncology Group (ECOG) score: 0-2 points, and life expectancy >3 months;
7. important organ function is acceptable, defined as: white blood cells ≥3.0×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥90g/L, glutamic pyruvic transaminase and glutamic oxalacetic transaminase ≤2.5 times the upper limit of normal value, serum creatinine < 178μmol/L;
8. voluntary participation and sign the informed consent.

Exclusion Criteria:

1. no suitable lesions for radiotherapy, or the limit of important organs at risk could not be met;
2. permanent discontinuation of PD-1/L1 inhibitors due to ≥ grade 3 immune-related toxic reactions;
3. serious cardiovascular or cerebrovascular diseases, severe liver or kidney dysfunction, serious and uncontrolled systemic infections or other contraindications, or any contraindications to radiotherapy, and some comorbidities should be re-evaluated after symptomatic treatment;
4. any active immune system disease or related history;
5. systemic immunosuppressive drugs are expected to be used during the study;
6. a history of severe uncontrollable central nervous system diseases or mental disorders, which may hinder the signing of informed consent or treatment compliance;
7. other important medical or physiological conditions (such as pregnancy or breastfeeding status);
8. patients who are known to be allergic to the drugs used in this study;
9. patients refuse or are unable to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | 6 weeks
  The proportion of treatment-related toxicities cases to the total evaluable cases, assessed according to CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
Objective response rate | 6 weeks
  Proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit.
Disease control rate | 6weeks
  Proportion of patients who achieved remission (PR+CR) or stable lesion (SD) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guangying Zhu, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Original research data including study protocol and statistical analysis plan will be shared after the study is completed and the research results are published.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available starting 6 months and ending 5 years following article publication.
Access Criteria: People who provide reasonable research protocols can get access to the data by contacting the researchers.